CLINICAL TRIAL: NCT01521286
Title: Population Based Surveillance to Estimate the Burden of Herpes Zoster and Postherpetic Neuralgia in Spain
Brief Title: Study to Estimate the Burden of Herpes Zoster and Postherpetic Neuralgia in Spain
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114617
Record Dates: First submitted 2012-01-26; First posted 2012-01-30 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Herpes Zoster
Keywords: Spain; cost; complications; incidence; adults; quality of life; Herpes Zoster; Surveillance
MeSH Terms: conditions — Herpes Zoster | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Group A: Subjects presenting with HZ episode.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — HZ and PHN booklet questionnaire and zoster brief pain inventory (ZBPI) questionnaire.

SUMMARY:
The purpose of this study is to collect data on the incidence, complications and impact on quality of life of herpes zoster (HZ) disease in adults >=50 years of age in Spain. This study will also collect data on costs related to the HZ disease, especially postherpetic neuralgia (PHN)

ELIGIBILITY:
Inclusion Criteria:

* A male or female >=50 years of age at the time of study enrolment presenting with acute HZ;
* HZ diagnosis for this HZ episode;

  * is the subject's first outpatient diagnosis; OR
  * took place at another site/ centre up to seven days before the initial visit for the present study;
* Ability to comply with study procedures*;
* Written informed consent obtained from the subject*. Note: * will be applicable to secondary objectives only and not for the primary objective to calculate incidence.

Exclusion Criteria:

• Subject participating in another research study. Note: This exclusion criteria is applicable to secondary objectives only and not for the primary objectives to calculate incidence.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult population, male or female, ≥50 years of age presenting with a HZ episode.
Sampling Method: Non-Probability Sample
Enrollment: 552 (Actual)
Dates: Start 2012-03; Primary Completion 2014-11 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Total number of HZ cases as recorded per participating practice, overall and within a specific age group and gender. | up to one year

SECONDARY OUTCOMES:
Occurrence of PHN, i.e. persistence of HZ-related pain. | 90, 180, and 270 days after onset of HZ.
Anamnestic information, clinical parameters and complications related to HZ. | Between Day 0 and Day 270
Direct medical, direct non-medical and indirect costs related to HZ. | Between Day 0 and Day 90
Pain assessment in HZ subjects. | At Day 90
Quality of life assessment in HZ subjects | Day 15, Day 30, Day 60 and Day 90
Direct medical, direct non-medical and indirect costs related to PHN. | At Day 90, Day 180 and Day 270
Pain assessment in PHN subjects. | At Day 90, Day 180 and Day 270
Quality of life assessment in PHN subjects. | At Day 90, Day 180 and Day 270

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Valencia

REFERENCES:
- [Derived] Diez-Domingo J, Curran D, Cambronero MDR, Garcia-Martinez JA, Matthews S. Economic Burden and Impact on Quality of Life of Herpes Zoster in Spanish Adults Aged 50 Years or Older: A Prospective Cohort Study. Adv Ther. 2021 Jun;38(6):3325-3341. doi: 10.1007/s12325-021-01717-7. Epub 2021 May 19. PMID 34013498